CLINICAL TRIAL: NCT01824355
Title: Performance of the Ninja 3 Plus Blood Glucose Monitoring System
Brief Title: Performance of an Investigational Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2012-010-01
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Monitoring System (Experimental): Untrained subjects with diabetes used the Ninja 3 PLUS Investigational BG Monitoring System. General enrollment criteria for the 'Intended Users' population:
  1. At least 60% of subjects were younger than 65 years of age.
  2. At least 20% had type 1 diabetes.
  3. At least 50% with type 2 diabetes were insulin users.
  Interventions: Device: Ninja 3 PLUS Investigational BG Monitoring System

INTERVENTIONS:
Device: Ninja 3 PLUS Investigational BG Monitoring System — Untrained subjects with diabetes performed self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the Ninja 3 PLUS Investigational BG Monitoring System. Study staff tested subject fingerstick blood. All BG results were compared to a reference laboratory glucose method.

SUMMARY:
The purpose of this study was to demonstrate that untrained subjects who have diabetes can operate the Investigational Blood Glucose Monitoring System (BGMS) and obtain valid glucose results.

ELIGIBILITY:
* Inclusion Criteria:

  1. Males and females, 18 years of age or older.
  2. People with type 1 or type 2 diabetes.
  3. Able to speak, read and understand English.
  4. Willing to complete all study procedures.
* Exclusion Criteria:

  1. Hemophilia or any other bleeding disorder.
  2. Pregnancy.
  3. Physical, visual or neurological impairments that would make the person unable to perform testing with the BGM.
  4. Previously participated in a blood glucose monitoring study using the Ninja 3 Plus BGMS.
  5. Working for a medical laboratory, hospital or other clinical setting that involves training on or clinical use of blood glucose meters.
  6. Working for a competitive medical device company, or having an immediate family member who works for such a company.
  7. A condition, which in the opinion of the investigator or designee, would put the person or study conduct at risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Caswell, PhD, Principal Investigator — Consumer Product Testing Co.
Locations (1):
- Consumer Product Testing Co., Fairfield, New Jersey, United States

REFERENCES:
- [Derived] Caswell M, Brown D, Frank J, Wallace JF, Pardo S. Accuracy and user performance evaluation of a blood glucose monitoring system which wirelessly transmits results to compatible insulin pumps. Curr Med Res Opin. 2020 May;36(5):757-764. doi: 10.1080/03007995.2020.1734919. Epub 2020 Mar 17. PMID 32096654

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the Monitoring System: Untrained subjects with diabetes used the Ninja 3 PLUS Investigational BG Monitoring System. General enrollment criteria for the 'Intended Users' population:
  1. At least 60% of subjects were younger than 65 years of age.
  2. At least 20% had type 1 diabetes.
  3. At least 50% with type 2 diabetes were insulin users.
  Ninja 3 PLUS Investigational BG Monitoring System: Untrained subjects with diabetes performed self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the Ninja 3 PLUS Investigational BG Monitoring System. Study staff tested subject fingerstick blood. All BG results were compared to a reference laboratory glucose method.
Period: Overall Study
Arm/Group | Intended Users of the Monitoring System
Started | 113
Completed | 110
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — unevaluable reference method results per | 1

BASELINE CHARACTERISTICS:
Population: All enrollees
Groups:
- Intended Users of the Monitoring System: Untrained subjects with diabetes used the Ninja 3 PLUS Investigational BG Monitoring System.
  Ninja 3 PLUS Investigational BG Monitoring System: Untrained subjects with diabetes performed self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the Ninja 3 PLUS Investigational BG Monitoring System. Study staff tested subject fingerstick blood. All BG results were compared to a reference laboratory glucose method.
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 113
Age, Customized [Mean (Full Range); unit: years]
  Age of enrolled subjects | 59.1 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 50
Race (NIH/OMB) [Number; unit: responses] — Subject responses could contain more than one race response, so number of responses will not equal number of participants.
  responses
    American Indian or Alaska Native | 1
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 26
    White | 84
    More than one race | 1
    Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 113

OUTCOME MEASURES:

1. Primary Outcome: Percent of Self Test Fingerstick Blood Glucose Results Within ±15 mg/dL (< 75 mg/dL) and Within ±20% (≥ 75 mg/dL) of the Laboratory Glucose Method
Description: Untrained subjects with diabetes who self-tested fingerstick blood used the Ninja 3 PLUS investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with capillary plasma BG results obtained with a reference laboratory glucose method - YSI Life Sciences (YSI) Analyzer. BG meter results were used to calculate the number of BGMS results within +/- 15mg/dL (for reference BG results <75mg/dL) and within +/- 20% (for reference BG results >=75mg/dL) of the YSI reference method results.
Time Frame: 1 hour
Population: 220 Blood Glucose results were analyzed. Each subject who completed (110 subjects) the study provided 2 Blood Glucose test results.
Measure: Number; unit: percentage of BG results
Units Other Than Participants: Blood Glucose Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 110
Number analyzed (Blood Glucose Results) | 220
percentage of BG results | 99.09

2. Secondary Outcome: Percent of Self Test Fingerstick Blood Glucose Results Within ±15 mg/dL (< 100 mg/dL) and Within ±15% (≥ 100 mg/dL) of the Laboratory Glucose Method
Description: Untrained subjects with diabetes who self-tested fingerstick blood used the Ninja 3 PLUS investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with capillary plasma BG results obtained with a reference laboratory glucose method - YSI Life Sciences (YSI) Analyzer. BG meter results were used to calculate the number of BGMS results within +/- 15mg/dL (for reference BG results <100mg/dL) and within +/- 15% (for reference BG results >=100mg/dL) of the YSI reference method results.
Time Frame: 1 hour
Population: as for outcome 1
Measure: Number; unit: percentage of Blood Glucose Results
Units Other Than Participants: Blood Glucose Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 110
Number analyzed (Blood Glucose Results) | 220
percentage of Blood Glucose Results | 97.73

3. Secondary Outcome: Percent of Self Test Fingerstick Blood Glucose Results Within ±12.5 mg/dL (< 100 mg/dL) and Within ±12.5% (≥ 100 mg/dL) of the Laboratory Glucose Method
Description: Untrained subjects with diabetes who self-tested fingerstick blood used the Ninja 3 PLUS investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with capillary plasma BG results obtained with a reference laboratory glucose method - YSI Life Sciences (YSI) Analyzer. BG meter results were used to calculate the number of BGMS results within +/- 12.5mg/dL (for reference BG results <100mg/dL) and within +/- 12.5% (for reference BG results >=100mg/dL) of the YSI reference method results.
Time Frame: 1 hour
Population: as for outcome 1
Measure: Number; unit: percentage of Blood Glucose Results
Units Other Than Participants: Blood Glucose Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 110
Number analyzed (Blood Glucose Results) | 220
percentage of Blood Glucose Results | 93.64

4. Secondary Outcome: Percent of Blood Glucose Results From Alternative Site Testing (AST) of the Palm Within ±15 mg/dL (< 75 mg/dL) and Within ±20% (≥ 75 mg/dL) of the Laboratory Method.
Description: Untrained subjects with diabetes self-tested Alternative Site (AST) Palm blood using the Ninja 3 PLUS investigational Blood Glucose Monitoring System (BGMS). BGMS AST results were compared with capillary plasma BG results obtained with a reference laboratory glucose method - YSI Life Sciences (YSI) Analyzer. BG meter results were used to calculate the number of AST BGMS results within +/- 15mg/dL (<75mg/dL YSI capillary plasma) and within +/- 15% (>=75mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 209 (220-11) Blood Glucose results were analyzed. 2 subjects had low blood sugar and per protocol their 4 AST BG results were not evaluable. 3 BG results were excluded as they were protocol deviations. One subject (2 BG results) did not complete testing within protocol timeframe and one subject (2 BG results) was unable to obtain AST blood.
Measure: Number; unit: percentage of AST Blood Glucose Results
Units Other Than Participants: Blood Glucose Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 110
Number analyzed (Blood Glucose Results) | 209
percentage of AST Blood Glucose Results | 97.13

5. Secondary Outcome: Percent of Fingerstick Blood Glucose Results Within ±15 mg/dL (< 75 mg/dL) and Within ±20% (≥ 75 mg/dL) of the Laboratory Glucose Method When Tested by Study Staff
Description: Study Staff tested subject fingerstick blood using the Ninja 3 PLUS investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with capillary plasma BG results obtained with a reference laboratory glucose method - YSI Life Sciences (YSI) Analyzer. BG meter results were used to calculate the number of BGMS results within +/- 15mg/dL (for reference BG results <75mg/dL) and within +/- 20% (for reference BG results >=75mg/dL) of the YSI reference method results.
Time Frame: one hour
Population: 220 Blood Glucose results were analyzed. Study Staff provided 2 Blood Glucose Test Results from each subject who completed (110 subjects) the study.
Measure: Number; unit: percentage of Blood Glucose Results
Units Other Than Participants: Blood Glucose Results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 110
Number analyzed (Blood Glucose Results) | 220
percentage of Blood Glucose Results | 100.0

6. Secondary Outcome: Number of Subject Responses That 'Strongly Agree' or 'Agree' or Are 'Neutral' With Questionnaire Statements
Description: Staff obtained subject responses using short questionnaires to provide feedback on instructions for use and the basic operation of the BGMS. Subjects could respond 'Strongly Agree' 'Agree' 'Neutral' 'Disagree' or 'Strongly Disagree.'
Time Frame: 1 hour
Population: Four subjects of those enrolled (113 subjects) had either missing or unevaluable questionnaire data.
Measure: Number; unit: participants
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 109
participants
  I find it easy to do a blood test with this meter | 108
  The meter display is easy to see and read | 108
  It was easy to understand my test results | 108
  I like the overall meter design | 106
  I find the meter easy to use | 106
  The instructions (User Guide) easy to understand | 105
  Instructions clearly explain how to run a test | 107
  Instructions clearly explain meter error messages | 108

ADVERSE EVENTS:
Time Frame: 1 hour subject visit
Arm/Group | Intended Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/113
Other Adverse Events (participants affected / at risk) | 3/113
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the Monitoring System (N=113)
Hypoglycemia (Endocrine disorders) | 1 (1)
Dizzy (Endocrine disorders) | 1 (1)
Headache (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days